CLINICAL TRIAL: NCT03296774
Title: Healthy Beyond Pregnancy: A Pilot Usability and Feasibility Trial
Brief Title: Healthy Beyond Pregnancy: Improving Postpartum Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO16090292
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2017-09

CONDITIONS: Postpartum Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Placebo Comparator): Usual postpartum care
  Interventions: Behavioral: Usual Care
- Healthy Beyond Pregnancy (Experimental): Web-based program for postpartum care and education and scheduling. Incentive for committing and returning for postpartum care.
  Interventions: Behavioral: Healthy Beyond Pregnancy

INTERVENTIONS:
Behavioral: Healthy Beyond Pregnancy — Web-based intervention grounded in behavioral economics and designed to improve adherence with postpartum care.
  Arms: Healthy Beyond Pregnancy
Behavioral: Usual Care
  Arms: Usual Care

SUMMARY:
Minority women and women of lower socioeconomic status are at significantly increased risk of unintended pregnancies, short inter-pregnancy interval, and short duration of breastfeeding. The consequences of poorly timed pregnancies and short duration of breastfeeding for the health of mothers, infants and children are well documented.

To decrease rates of poorly timed pregnancies, increase breastfeeding duration and address other postpartum concerns women must be engaged in their postpartum care outside of the traditional postpartum visit. In addition to contraceptive counseling and breastfeeding support, providers discuss a number of important maternal and child health issues at the postpartum visit. These include (1) screening and referral for postpartum mood disorders (2) screening for cardiometabolic consequences of pregnancy complications, (3) discussing inter-conception care and (4) connecting women with a primary care provider. Thus, as recommended by numerous professional societies, the standard postpartum visit at 4 to 6 weeks after delivery has considerable value to women's postpartum care.

Attendance rates for the postpartum visit are markedly lower for women with limited resources contributing to racial and economic health disparities. Despite receiving excellent prenatal care, only 40% of the economically disadvantaged women who receive prenatal care at the Magee outpatient clinic return for their postpartum visit. These parallel national trends, where 60% of women with Medicaid insurance return for a postpartum checkup compared with over 82% of women with private insurance. Medicaid programs serve pregnant women who are particularly vulnerable to poor health outcomes and thus this gap is critical. Additionally, minority women disproportionally receive Medicaid and thus interventions that focus on Medicaid recipients have the potential to address racial as well as economic disparities. These data demonstrate that the current care model does not engage all women to make good health care decision postpartum and is disproportionately failing our most vulnerable moms and babies.

Empirically derived concepts from behavioral economics can be leveraged to design interventions that support participants to make better health decisions and may be particularly useful for postpartum care.

The feasibility trial will focus on four tenants of behavioral economics-bounded rationality (information overload), status quo bias (lack of self-control), hovering (limited attention), and framed incentives-- that have been successfully used to tackle stubborn health problems such as smoking and obesity. Importantly, unlike tobacco cessation or weight loss, many aspects of postpartum care such as compliance with the visit or uptake of LARC, do not require on-going action on part of the patient and thus may be particularly amenable to the lessons of behavioral economics.

Specific Aim 1: To conduct a pilot trial evaluating the feasibility and acceptability of a future randomized trial to determine the efficacy of Healthy Beyond Pregnancy on adherence with the postpartum visit.

Specific Aim 2: To determine the impact of Healthy Beyond Pregnancy on adherence with the postpartum visit.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum 6-72 hours from delivery, aged 18-50, receipt of prenatal care through the Magee-Womens Hospital outpatient clinic and UPMC for You Medicaid insurance.

Exclusion Criteria:

* Delivery less than 24 weeks, fetal or neonatal death, non-English speaking, no text-enabled phone

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy based study
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Number of eligible participants who consent and complete study intervention | 1-4 days postpartum
  Assess the feasibility of a larger randomized controlled trial

SECONDARY OUTCOMES:
Adherence with postpartum visit- number of participants who return for postpartum visit. | 21-56 days after delivery
  Did participant come for postpartum visit

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Himes KP, Donovan H, Wang S, Weaver C, Grove JR, Facco FL. Healthy Beyond Pregnancy, a Web-Based Intervention to Improve Adherence to Postpartum Care: Randomized Controlled Feasibility Trial. JMIR Hum Factors. 2017 Oct 10;4(4):e26. doi: 10.2196/humanfactors.7964. PMID 29017990